CLINICAL TRIAL: NCT06423313
Title: The Comparison of Total Intravenous Anesthesia and Inhalation Anesthesia Effects on Postoperative Recovery by Quality of Recovery (QoR-40) in Septorhinoplasty
Brief Title: Effects of Anesthesia Type on QoR-40
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2024/07-1
Record Dates: First submitted 2024-05-03; First posted 2024-05-21 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: General Anesthesia; İnhalation Anesthetics; Quality of Recovery
Keywords: total intravenous anesthesia; anesthesia maintenance; inhalation anesthesia; quality of recovery-40

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group TIVA
  Interventions: Procedure: maintenance of anesthesia
- Group Inhalation
  Interventions: Procedure: maintenance of anesthesia

INTERVENTIONS:
Procedure: maintenance of anesthesia — Types used to maintain anesthesia

SUMMARY:
To compare the effects of total intravenous anesthesia and inhalation anesthesia used for maintenance on postoperative recovery in patients undergoing septorhinoplasty surgery under general anesthesia, using the recovery quality score (QoR-40).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA I-II-III risk group
* Patients whose consent was obtained with an informed consent form
* Patients who will undergo septorhinoplasty surgery

Exclusion Criteria:

* -ASA >3
* Psychiatric illness that prevents them from answering the questionnaire
* Patients with a history of chronic opioid and benzodiazepine use as it may affect recovery time
* Severe renal and hepatic insufficiency
* Severe respiratory and cardiovascular disease
* Patients with a body mass index >30 kg m2
* Patients with a known history of allergy or contraindication to any of the drugs to be used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include intubated patients who will undergo septorhinoplasty surgery under general anesthesia, aged 18-65 years, in the American Society of Anesthesiology (ASA) I-II-III risk class.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
quality of recovery-40 questionnaire | up to 24 hour after surgery
  measurement of recovery quality in the first 24 hours after extubation with quality of recovery-40 questionnaire. Quality of recovery-40 questionnaire scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

SECONDARY OUTCOMES:
postoperative complications | up to 24 hour after surgery
  complications that may occur in the postoperative period
duration of extubation | end of the surgery
  time between the last suture and extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No